CLINICAL TRIAL: NCT02825511
Title: Assessment of the Clinic-pathological Correlation of Basal Cell Carcinoma: Establishment of a Prospective Observational Cohort and Followed 3 Years
Brief Title: Assessment of the Clinic-pathological Correlation of Basal Cell Carcinoma
Acronym: CAC-CBC
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/18
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma, histological diagnosis, prognostic impact
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A cohort of basal cell carcinoma: A cohort of surgically treated BCC, primitive clinically suspected or previously biopsied on a 4-month period, an expected number of 3 200 cases. The management of the BCC will be consistent with current recommendations. BCC recurrence and those who received prior medical treatment will be excluded.

SUMMARY:
Assessment of the concordance of the initial clinical and histological diagnosis and to explore its prognostic impact in terms of risk of recurrence.

DETAILED DESCRIPTION:
The skin cancer is a major public health problem whose incidence is increasing due to the aging population. Among them, basal cell carcinoma (BCC) is a daily concern the dermatologist. The recommendation of good practice for the BCC of support has been established according to French agency methodology in 2004 : "Agence Nationale d'Accréditation et d'Evaluation en Santé" (ANAES). This classification is based on clinical and pathological use of sometimes mismatched terminology pretending to clinical reality with discrepancies between the clinical appearance and histology. On the other hand the simplified classification of recommendations has never been tested and validated on a large series of BCC. Probabilistic margins applied based on clinical assessment of clinical and pathological subtype, it seems interesting to evaluate the consistency of the initial clinical diagnosis and histological diagnosis and to explore its prognostic impact in terms of risk of recurrence.

This study could lead to improved clinical and pathological classification and allow amending the current recommendations of the surgical management of the BCC.

ELIGIBILITY:
Inclusion Criteria:

* Primitive BCC
* BCC clinically suspected or previously biopsied
* Supports conventional surgical or micrographic techniques.
* Patient able to sign a consent after reading the briefing note

Exclusion Criteria:

* Recurrent CBC
* prior medical treatment
* BCC assigned to another operator for removal
* Genodermatosis underlying (xeroderma pigmentosum - Gorlin syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BCC primitive, clinically suspected or previously biopsied
Sampling Method: Non-Probability Sample
Enrollment: 2738 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Dimension of basal cell carcinoma. | Day 1
Number of clinical type of basal cell carcinoma (nodular, superficial or sclerodermiform) | Day 1
Number of histological type of basal cell carcinoma (nodular, superficial, infiltrating or sclerodermiform) | Day 1

SECONDARY OUTCOMES:
Number of the disease according to region (head, leg, arm, eyelid, lip,...) | Day 1
Clinical aggressiveness Score with "Agence Nationale d'Accréditation et d'Evaluation en Santé" (ANAES) criteria | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel AMICI, MD, Principal Investigator — University Hospital, Bordeaux
Locations (17):
- France (17):
  - Wiart (Dermatologue - Armentieres), Armentières
  - Dupin (Dermatologue - Auch), Auch
  - University Hospital of Bordeaux - Hospital Saint André, Bordeaux
  - Will (Dermatologue - Brumath), Brumath
  - Ruto (Dermatologue - Evreux), Évreux
  - Jacquet (Dermatologue - Hyeres), Hyères
  - Tranchand (Dermatologue - Le Puy En Velay), Le Puy-en-Velay
  - Groupe Hospitalier de L'Institut Catholique de Lille, Lille
  - Bacconier (Dermatologue - Marseille), Marseille
  - Haberstroh (Dermatologue - Mulhouse), Mulhouse
  - Bolzinger (Dermatologue - Nay), Nay
  - CHU de Nice, Nice
  - Chaussade (Dermatologue - Paris), Paris
  - Tanguy (Dermatologue - Pau), Pau
  - Bailly (Dermatologue - Toulouse), Toulouse
  - Chu de Toulouse, Toulouse
  - Lulin (Dermatologue - Vendome), Vendôme

IPD SHARING:
Plan to Share IPD: No